CLINICAL TRIAL: NCT00224562
Title: The RATIO Registry: French Registry on Opportunistic and Severe Bacterial Infections and Lymphoma in Patients Treated With TNF-a Antagonists
Brief Title: The RATIO: Registry of Infections and Lymphoma in Patients Treated With TNF-a Antagonists
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Other Study IDs: 1; INSERM
Record Dates: First submitted 2005-09-14; First posted 2005-09-23 (Estimated); Last update posted 2005-10-26 (Estimated); Status verified 2004-02

CONDITIONS: Rheumatoid Arthritis; Crohn's Disease; Ankylosing Spondylitis; Psoriasis
Keywords: TNF alpha antagonists; infections; lymphoma; safety
MeSH Terms: conditions — Arthritis, Rheumatoid; Crohn Disease; Spondylitis, Ankylosing; Psoriasis; Infections; Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Drug: TNF-alpha antagonists

SUMMARY:
The RATIO registry is a French registry designed by a multidisciplinary group to collect data on opportunistic and severe bacterial infections and lymphoma in patients treated with TNF-a antagonists ( infliximab, etanercept and adalimumab). A total of 486 medical units in metropolitan France participate in the RATIO registry. All diagnosis are retained after validation by 2 qualified infectious disease or haematologist physicians (on the basis of the standardized case report form, the hospitalisation summary, and the microbiological and radiological results). Risk factors for developing these conditions when treated by TNF-a antagonists will be identified in a case control study. Incidence of these diseases will be calculated.

ELIGIBILITY:
Inclusion Criteria for cases:

* past or current treatement with TNF-a antagonists
* either lymphoma severe bacterial infection opportunistic infection

Inclusion Criteria for controls:

* matched with cases by gender, age (+/- 5 years), underlying disease (rheumatoid arthritis, ankylosing spondylitis, Crohn's disease, or psoriasis)
* past or current treatement with TNF-a antagonists
* no lymphoma, severe bacterial infection, opportunistic infection (same as case)

Exclusion Criteria:

* none

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-02

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Mariette, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Dominique Salmon, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Marc Lemann, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- All French departments of rheumatology, internal medicine, gastro-enterology, dermatology, infectious diseases, intensive care unit, oncology and haematology, paediatrics and chest medicine, All Cities, France

REFERENCES:
- [Derived] Lanternier F, Tubach F, Ravaud P, Salmon D, Dellamonica P, Bretagne S, Couret M, Bouvard B, Debandt M, Gueit I, Gendre JP, Leone J, Nicolas N, Che D, Mariette X, Lortholary O; Research Axed on Tolerance of Biotherapies Group. Incidence and risk factors of Legionella pneumophila pneumonia during anti-tumor necrosis factor therapy: a prospective French study. Chest. 2013 Sep;144(3):990-998. doi: 10.1378/chest.12-2820. PMID 23744173
- [Derived] Tubach F, Salmon D, Ravaud P, Allanore Y, Goupille P, Breban M, Pallot-Prades B, Pouplin S, Sacchi A, Chichemanian RM, Bretagne S, Emilie D, Lemann M, Lortholary O, Mariette X; Research Axed on Tolerance of Biotherapies Group. Risk of tuberculosis is higher with anti-tumor necrosis factor monoclonal antibody therapy than with soluble tumor necrosis factor receptor therapy: The three-year prospective French Research Axed on Tolerance of Biotherapies registry. Arthritis Rheum. 2009 Jul;60(7):1884-94. doi: 10.1002/art.24632. PMID 19565495